CLINICAL TRIAL: NCT06182826
Title: Effect of Core Engagement Exercises and Routine Exercise Therapy on Low Back Pain in Middle School Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/24
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a single blinded randomized controlled trial having two groups. One group will be given Core Stabilization Protocol along with Routine exercise therapy whereas other group will only receive Routine Exercise therapy protocol. Both groups will be recruited concurrently.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients in this group will receive Core Stability Protocol with Routine Exercise Protocol. A total of 3 sessions per week for 6 weeks will be given.
  Interventions: Procedure: Core Stability protocol; Procedure: Routine exercise therapy
- Group B (Active Comparator): Patients will receive Routine Exercise Protocol. A total of 3 sessions per week for 6 weeks will be given.
  Interventions: Procedure: Routine exercise therapy

INTERVENTIONS:
Procedure: Core Stability protocol — 5 Minutes Warm up Hamstring stretch Back Extensor Stretch Hip Flexor Stretch Jumping Rope Stair Stepping Mountain Climbers Curl Up Side Planks Bird Dog Frequency: 3 sessions per week for six weeks. Time Duration: Approx. 30 to 45 minutes
  Arms: Group A
Procedure: Routine exercise therapy — 5 Minutes Warm up Hamstring stretch Back Extensor Stretch Hip Flexor Stretch Jumping Rope Stair Stepping Mountain Climbers Frequency: 3 sessions per week for six weeks. Time Duration: Approx. 30 to 45 minutes

SUMMARY:
Low back pain is defined as the region of pain between the lower ribs and hips. Low back pain with respect to middle school children corresponds to the age where children and adolescents go to school for longer periods of time, having heavy bags, assuming poor postures while sitting for prolonged hours. Poor posture, prolonged sitting and lack of physical activity results in back pain that leads to poor performance in school as well as attendance.

DETAILED DESCRIPTION:
Middle school children are the children of the age where they spend most of their hours sitting in school. Low back pain often goes undiagnosed and unreported in children which persists and if left untreated, causes problems in later stages in life.

Low back pain is the region of pain from lower ribs to hips. Children and teenagers often have lower back discomfort, which may be brought on by several conditions, including poor lifting skills, bad posture, and overuse injuries from sports or other physical activity. According to estimates, up to 50% of school-aged children may sometimes have lower back discomfort. The muscles that surround our spine are considered the "core" of our body. It is composed of the abdominal muscles on your front and sides, the erector muscles and gluteus. Each and every one of these muscles must work together in order to enhance the stability of the spine. When muscles contract they create force and stiffness. It is the stiffness part that is important for stability. When the core fails to meet the stability demands placed on the body during a certain lift, parts of the spine will be overloaded with forces that increase injury risk and performance will suffer. For that, various warm up exercises, stretches and mobility exercises are performed so that the body can work as stable linked system that works efficiently as well.

ELIGIBILITY:
Inclusion Criteria:

* Middle aged school children between age 9 and 14.
* Both male and female.
* Back pain of 2 or greater on NPRS

Exclusion Criteria:

* Structural observational deformity (kyposis, lordosis, scoliosis)
* History of post spinal surgery
* Acute low back pain flare up
* Pain or any other injury of lower limbs

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 6 week
  Pain will be measured using the Numeric Pain Rating Scale, which is an 11-item scale.
Trunk Extensor Endurance | 6 week
  Trunk extensor endurance will be measured using McGill Endurance Test Battery
Trunk Flexor Endurance | 06 Week
  Trunk flexor endurance will be measured using McGill Endurance Test Battery
Lateral Endurance | 06 Week
  Trunk lateral endurance will be measured using McGill Endurance Test Battery

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan